CLINICAL TRIAL: NCT05380869
Title: Point-of-care Procalcitonin Testing for Lower Respiratory Tract Infection in Outpatient Care
Brief Title: POCT PCT in Outpatient LRTI
Acronym: POCT-PCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8736_MPG_23b2019
Record Dates: First submitted 2022-04-12; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: Antimicrobial Stewardship; Exacerbation of Allergic Asthma; Exacerbation Copd; Community-acquired Pneumonia; Lower Respiratory Tract and Lung Infections
Keywords: Procalcitonin; Point-of-care-Testing; Antimicrobial stewardship
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: Diagnostic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Point-of-care test Procalcitonin for LRTI (Other): Diagnostic study, a POCT-PCT is done in all included patients
  Interventions: Diagnostic Test: Point-of-care Test

INTERVENTIONS:
Diagnostic Test: Point-of-care Test — to test Point-of-care procalcitonin in suspected pneumonia

SUMMARY:
Lower respiratory tract infections (LRTI) in patients with chronic lung diseases are a common acute reason to consult respiratory practitioners and often lead to inadequate prescription of antibiotics. The primary objective of the investigators study was to determine the diagnostic accuracy of point-of-care testing (POCT) for procalcitonin (PCT) in identifying pneumonia as a bacterial infection in outpatients with LRTI.

DETAILED DESCRIPTION:
Lower respiratory tract infections (LRTI) are a common acute reason to consult general practitioners or lung specialists and most patients receive an antibiotic prescription. Despite the vast majority of LRTI are caused by viruses, the lack of clinical, radiological, and laboratory tests to safely rule out bacterial involvement in LRTI still drives antibiotic treatment today Procalcitonin (PCT) has been shown to be a useful biomarker for differentiating between viral and bacterial infections in the emergency department and is now available as a point-of-care testing (POCT). The primary objective of the investigators study was to determine the diagnostic accuracy of POCT PCT in identifying bacterial infection in outpatients with LRTI. All patients aged 18 years or older with signs and symptoms of an LRTI as the leading diagnosis of the respiratory physicians are eligible. The medical assistant measure PCT from venous or capillary whole blood using the portable commercially available BRAHMS PCT direct point-of-care test (Thermo-Fischer Scientific). The stepwise procedure involve pipetting 20µl of the sample into the test disc before loading this onto the analyzer and pressing run. This immunoassay provides a quantitative result in 20 minutes. In suspicion of pneumonia (positive auscultation finding or clinical noticed symptoms compatible with pneumonia) a chest x-ray will be done. Members of the study team conduct standardised phone interviews of all participants on day 28.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical diagnosis of lower respiratory tract infection

Exclusion Criteria:

* Active malignancies
* Cystic fibrosis
* Solid organ or stem cell transplantation
* Chronic infection (endocarditis, osteomyelitis, active tuberculosis)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Description of outpatients with lower respiratory tract infection | up to 5 weeks
  The study population will be described in terms of demographic characteristics using descriptive statistics.
Determining the diagnostic accuracy of POCT PCT in identifying bacterial infection in outpatients with LRTI using portable commercially available BRAHMS PCT direct point-of-care test. | up to 5 weeks
  For the diagnostic accuracy of the PCT the receiver operating characteristic (ROC) curves and the area under the curve (AUC) will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School Hannover, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No